CLINICAL TRIAL: NCT00002239
Title: A Controlled Phase 2 Trial Assessing Three Doses of T-20 in Combination With Abacavir, Amprenavir, Ritonavir, and Efavirenz in HIV-1 Infected Adults
Brief Title: A Study to Compare Three Doses of T-20 When Given in Combination With Abacavir, Amprenavir, Ritonavir, and Efavirenz to HIV-Infected Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Trimeris (Industry)
Purpose: Treatment
Other Study IDs: T20-206; 295B
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-11-15 (Estimated); Status verified 2005-11

CONDITIONS: HIV Infections
Keywords: HIV-1; Dose-Response Relationship, Drug; Drug Therapy, Combination; VX 478; Anti-HIV Agents; pentafuside; abacavir; efavirenz
MeSH Terms: conditions — HIV Infections | interventions — Enfuvirtide; Ritonavir; abacavir; amprenavir; efavirenz

INTERVENTIONS:
Drug: Enfuvirtide
Drug: Ritonavir
Drug: Abacavir sulfate
Drug: Amprenavir
Drug: Efavirenz

SUMMARY:
The purpose of this study is to see if it is safe and effective to give T-20, a new type of anti-HIV drug, with a combination of other anti-HIV drugs. The other anti-HIV drugs used are abacavir (ABC), amprenavir (APV), ritonavir (RTV), and efavirenz (EFV). Three different doses of T-20 are tested.

DETAILED DESCRIPTION:
Patients are assigned to one of four groups. Three dose groups receive a background antiretroviral regimen (ABC, APV, RTV, and EFV) and T-20, which is given at one of three doses on a twice-daily regimen. The fourth group (control) receives the background antiretroviral regimen alone. For each treatment group, 17 patients are enrolled. Treatment is administered for 16 weeks, followed by a 32-week treatment extension, and a 2-week follow-up period. The following are assessed throughout the trial: safety parameters (as measured by hematology, clinical chemistry, urinalysis, and treatment-emergent adverse events); virologic and immunologic activity; phenotypic and genotypic resistance; T-20 plasma levels; and pharmacokinetics of T-20 and oral antiretrovirals. The total study duration is 1 year.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-positive.
* Have an HIV level (viral load) between 400 and 100,000 copies/ml at the screening visit.
* Have taken at least 1 PI (protease inhibitor) for at least 16 weeks, and have had no interruptions in their most recent PI-containing anti-HIV drug regimen.
* Are at least 18 years old.
* Agree to abstinence or use of 2 effective methods of birth control, including a barrier method, during the study.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have ever taken an NNRTI (nonnucleoside reverse transcriptase inhibitor).
* Have an opportunistic (HIV-related) infection.
* Have had an unexplained fever of at least 38.5 C for 7 days in a row within 30 days prior to screening.
* Have had diarrhea lasting at least 15 days within 30 days prior to screening.
* Have ever taken abacavir, amprenavir, or efavirenz (ABC, APV, or EFV).
* Have certain genetic characteristics (drug resistance mutations) that could change the way a drug acts in the body.
* Are allergic to any of the study medications.
* Have a tumor other than certain skin or cervical cancers.
* Are on chemotherapy that cannot be discontinued during the study.
* Are taking an investigational drug within 30 days prior to screening.
* Have ever received an HIV vaccine.
* Are taking certain medications.
* Abuse drugs or alcohol.
* Have hemophilia or another blood clotting disorder.
* Have had an organ transplant.
* Are pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68
Dates: Start 1999-05

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Pacific Oaks Research, Beverly Hills, California
  - UCLA Care Ctr, Los Angeles, California
  - ViRx Inc, Palm Springs, California
  - Donald Northfelt, Palm Springs, California
  - UCSD, San Diego, California
  - ViRx Inc, San Francisco, California
  - Quest Clinical Research, San Francisco, California
  - Dupont Circle Physicians Group, Washington D.C., District of Columbia
  - IDC Research Initiative, Altamonte Springs, Florida
  - Gary Richmond MD, Fort Lauderdale, Florida
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Washington Univ School of Medicine, St Louis, Missouri
  - New York Univ Med Ctr, New York, New York
  - Trimeris Inc, Durham, North Carolina
  - Associates of Med and Mental Health, Tulsa, Oklahoma
  - Pennsylvania Oncology and Hematology Associates, Philadelphia, Pennsylvania
  - Philadelphia FIGHT, Philadelphia, Pennsylvania
  - Univ of Pittsburgh, Pittsburgh, Pennsylvania
  - Central Texas Clinical Research, Austin, Texas